CLINICAL TRIAL: NCT03395041
Title: Periodontal Disease, Inflammation and Atherosclerosis Progression in Patients With Acute Coronary Syndromes - the ATHERODENT Study
Brief Title: Periodontal Disease, Inflammation and Acute Coronary Syndromes
Acronym: ATHERODENT
Status: Completed | Type: Observational
Sponsor: Cardio Med Medical Center (Industry)
Collaborators: University of Targu Mures, Romania (Other); University Hospital of Targu Mures, Romania (Other)
Responsible Party: Sponsor
Other Study IDs: CM0117-ATD
Record Dates: First submitted 2018-01-03; First posted 2018-01-10 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2019-07

CONDITIONS: Coronary Stenosis; Periodontal Diseases; Acute Coronary Syndrome; Non-ST Elevation Myocardial Infarction; Unstable Angina; Acute Myocardial Infarction; Atherosclerosis; Atheromatous Plaques
Keywords: vulnerable plaque, CT imaging, oral bacteria, inflammation
MeSH Terms: conditions — Coronary Stenosis; Periodontal Diseases; Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; Angina, Unstable; Atherosclerosis; Plaque, Atherosclerotic; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for determination of miRNA fractions associated with coronary plaque vulnerability
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATD - SG 01: Patients with acute coronary syndrome in whom dental examination performed in the first 7 days after the index event revealed the presence of periodontal disease.
  They will undergo complex cardiac imaging tests to assess plaque vulnerability and severity of coronary artery disease.
  Interventions: Diagnostic Test: cardiac imaging tests
- ATD - SG 02: Patients with acute coronary syndrome in whom dental examination performed in the first 7 days after the index event did not reveal the presence of periodontal disease.
  They will undergo complex cardiac imaging tests to assess plaque vulnerability and severity of coronary artery disease.
  Interventions: Diagnostic Test: cardiac imaging tests

INTERVENTIONS:
Diagnostic Test: cardiac imaging tests — cardiac computed tomography, echocardiography, intravascular ultrasound, optical coherence tomography

SUMMARY:
Recent studies have shown that the systemic inflammation caused by periodontal disease (PD) can determine important changes in the coronary arteries, favoring atherosclerosis progression and development of acute coronary syndromes (ACS). The aim of ATHERODENT study is to assess the interrelation between PD, inflammation and progression of coronary atherosclerosis in patients with ACS. Material and methods: This case-control observational study will enroll 100 patients (group 1 - ACS and associated PD, and group 2 -ACS and no PD), in whom the following data will be collected: (1) demographic and clinical data, (2) cardiovascular risk factors, (3) full characterization of PD markers, (4) systemic inflammatory biomarkers, (5) imaging biomarkers derived from transthoracic echocardiography, computed tomography, coronary angiography, optical coherence tomography and intravascular ultrasound, and (6) assessment of the presence of specific oral bacteria in samples of coronary plaques collected by coronary atherectomy, which will be performed during percutaneous revascularization interventions, when indicated in selected cases, in the atherectomy sub-study. The follow-up will be performed at 1, 3, 6, 12, 15, 18 and 24 months. The primary endpoint of the study will be represented by the rate of major adverse cardiovascular events (MACE rates) in PD vs non-PD patients and in correlation with: (1) the level of systemic inflammation triggered by PD and/or by ACS at baseline; (2) the vulnerability degree of atheromatous plaques in the coronary tree (culprit and non-culprit lesions); and (3) the presence and burden of oral bacteria in atheromatous plaques. Secondary endpoints will be represented by: (1) the rate of progression of vulnerability degree of non-culprit coronary plaques; (2) the rate of progression of atheromatous burden and calcium scoring of the coronary tree; and (3) the rate of occurrence of left ventricular remodeling and postinfarction heart failure.

DETAILED DESCRIPTION:
ATHERODENT is a case-controlled observational clinical study, conducted in two clinical sites: University of Medicine and Pharmacy Tirgu Mures, Romania, and Cardio Med Medical Center - Laboratory of Advanced Research in Multimodality Imaging.

The primary objective of ATHERODENT is to assess the interrelation between PD, inflammation and atherosclerosis progression in patients who suffered an ACS and have concomitant PD vs those with ACS and no PD, using (1) invasive and non-invasive imaging techniques for characterization of vulnerable coronary plaques; (2) full characterization of PD; and (3) complex assessment of systemic vulnerability based on systemic inflammation-related biomarkers.

The secondary objectives of ATHERODENT are:

1. to study the correlation between PD and coronary plaque vulnerability
2. to assess the correlation between PD and severity of coronary atherosclerosis
3. to assess the presence and burden of oral bacteria in coronary atheromatous plaques collected during atherectomy and their relation with plaque vulnerability and evolution following an ACS (in the atherectomy sub-study).

Baseline will be considered as the moment of the index event and related hospitalization. The index event will be considered the ACS and patients will be randomized in the study at maximum 7 days post ACS. The follow-up visits will be performed at 1, 3, 6, 12, 15, 18 and 24 months after randomization.

The following procedures will be performed at baseline:

1. recording of demographic and clinical data (age, gender, personal history)
2. determination of serum lipids, blood counts, glycemia, urea, creatinine, liver enzymes
3. determination of the biomarkers expressing the severity of the acute coronary syndrome and heart damage (hs-Troponin, NT-proBNP)
4. determination of serum levels inflammatory biomarkers and adhesion molecules at the moment of the index event (hs-CRP, matrix metalloprotease, interleukin-6, VCAM, ICAM)
5. determination of specific micro-RNAs related to plaque vulnerability
6. echocardiography (+ speckle tracking) for assessment of left ventricular function and size
7. full characterization of PD (dental plaque/tartar, gingival retraction, gingival bleeding, etc.)
8. microbiological determination of oral bacteria from the periodontal pockets
9. non-invasive imaging by coronary angioCT for all the coronary tree and characterization of vulnerability markers and atherosclerosis severity, using surrogate imaging biomarkers such as calcium score, necrotic core, plaque burden, low density atheroma, positive remodeling, epicardial fat volume
10. invasive imaging performed during invasive revascularization procedures, using intracoronary imaging techniques (OCT, IVUS) and quantification of invasive imaging biomarkers in culprit and non-culprit lesions, such as macrophage content, thickness of fibrous cap and necrotic core.
11. atherectomy of coronary culprit atheromatous plaques (in the atherectomy sub-study), performed during the revascularization procedure when indicated, in selected cases, followed by histological examination of the samples collected in order to identify specific antigens related to oral microbiota in the atheromatous tissue of coronary vulnerable plaques.

Follow-up will be performed at 1, 3, 6, 12, 15, 18 and 24 months after randomization, including assessment of clinical data, echocardiography and registration of MACE and adverse events.

In addition, complex imaging assessment using Angio CT will be performed at 2 years to assess atherosclerosis progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years;
* Patients who have signed the written informed consent;
* Patients with ACS (unstable angina or non-ST segment elevation myocardial infarction) occurring with maximum 7 days prior to enrollment

Exclusion Criteria:

* Patient's refusal to participate in the study;
* Sensitivity to the contrast substance;
* Women of reproductive age who do not use contraceptive methods;
* Pregnant women;
* Any malignancy within the last 5 years;
* Any disease or comorbidity that can reduce life expectancy to less than 2 years;
* Acute or chronic renal failure;
* Non-compliant patients who, in the opinion of the investigators, will not present to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndromes (unstable angina or NSTEMI), who undergo invasive coronary angiography +/- revascularization (according to local protocols).
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
The rate of major adverse cardiovascular events (MACE rates). | 24 months
  Cardiac death, need for target vessel revascularization (with target vessel defined as the vessel with a vulnerable plaque), or reinfarction.

SECONDARY OUTCOMES:
The rate of progression of vulnerability degree of non-culprit coronary plaques | 24 months
  Increased severity in vulnerability indexes determined by cardiac imaging tests in the coronary tree
The rate of progression of atheromatous burden and calcium scoring | 24 months
  Increase in atheromatous plaque burden and calcium scoring of the entire coronary tree as determined by Cardio CT
The occurrence of left ventricular remodeling and post-infarction heart failure | 24 months
  Development of ventricular remodeling defined as increase in ventricular diameters with>15% compared to baseline, and of post-infarction heart failure, defined as left ventricular ejection fraction <45% in the posti-infarction period

CONTACTS AND LOCATIONS:
Overall Officials: Theodora Benedek, Prof, Principal Investigator — University of Medicine and Pharmacy Tirgu Mures, CardioMed Medical Center
Locations (1):
- Cardio Med, Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available to other researchers from the same group and to other collaborating groups and can be used for further statistical sub-analysis
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available immediately after completion of the enrolment and will remain available for at least 5 years.